CLINICAL TRIAL: NCT00228059
Title: A 52-week, Open-label Extension Study to Evaluate the Safety and Tolerability of Licarbazepine 750- 2000 mg/Day in the Treatment of Manic Episodes of Bipolar I Disorder
Brief Title: An Open-label Extension Study to Evaluate the Safety and Tolerability of Licarbazepine in the Treatment of Manic Episodes of Bipolar I Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC477D2301E1
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar disorder, manic episode/treatment/licarbazepine
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
This extension study is designed to investigate the long-term safety and tolerability of licarbazepine 750-2000 mg/day over 52 weeks in patients who completed the 3-week double-blind study CLIC477D2301.

DETAILED DESCRIPTION:
A 52-week, open-label extension study to evaluate the safety and tolerability of licarbazepine 750- 2000 mg/day in the treatment of manic episodes of bipolar I disorder

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent provided prior to participation in the extension study
2. successful completion of study CLIC477D2301
3. willingness and ability to comply with all study requirements

Exclusion Criteria:

1. premature discontinuation from study CLIC477D2301
2. failure to comply with the study CLIC477D2301 protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of licarbazepine with respect to adverse events, serious adverse events, changes in laboratory values, ECGs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmcuticals, Study Chair — Novartis
Locations (1):
- Investigational Site, Cerritos, California, United States

REFERENCES:
- See also: (Click here for further information and to find an investigational site near you) — http://www.novartisclinicaltrials.com/etrials/DiseaseID10/Bipolar-Disorder-clinical-trials.go